CLINICAL TRIAL: NCT04287933
Title: Role of Drain in Decreasing Postoperative Complications After Cesarean Section
Brief Title: Role of Drain in Decreasing Postoperative Complications
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aljazeera Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: drain
Record Dates: First submitted 2020-02-26; First posted 2020-02-27 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Cesarean Section Complications

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drain (Active Comparator)
  Interventions: Device: Drain insertion
- No drain (No Intervention)

INTERVENTIONS:
Device: Drain insertion — insertion of a drain
  Arms: Drain

SUMMARY:
postoperative complications are common after cesarean section

DETAILED DESCRIPTION:
wound infection can occur after cesarean section

ELIGIBILITY:
Inclusion Criteria:

Women undergoing cesarean section

Exclusion Criteria:

* Women who deliver by normal vaginal delivery

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women who will have complications after cesarean sectin
Enrollment: 200 (Estimated)
Dates: Start 2020-03-02 (Estimated); Primary Completion 2020-07-03 (Estimated); Study Completion 2020-08-10 (Estimated)

PRIMARY OUTCOMES:
The number of women who will have complications | within 2 weeks
  How many women who will have complications postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, PhD, Study Chair — Algezeera hospitaland National Research Centre ,Egypt
Locations (1):
- Algazeerah, Giza, Egypt